CLINICAL TRIAL: NCT00140673
Title: A Placebo-controlled, Multi-country & Multi-center Study to Assess the Efficacy, Safety & Immunogenicity of 2 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Infants
Brief Title: A Study to Test 2 Doses of the HRV Vaccine in Healthy Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 444563/023
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: Rotavirus

SUMMARY:
The main objectives of this study are: 1) In a subset (N = 20 000), to determine vaccine efficacy against severe rotavirus (RV) gastroenteritis (GE) during the period starting from 2 weeks after Dose 2 until one year of age. 2) In all subjects (N = 60 000), to determine the safety of GSK Biologicals' HRV vaccine with respect to definite intussusception (IS) within 31 days (Day 0-Day 30) after each HRV vaccine dose.

DETAILED DESCRIPTION:
The study has two groups: Group HRV and Group Placebo. Two oral doses administered to healthy infants who are 6-13 weeks of age at the time of Dose 1, according to a 0, 1 to 2-month schedule. Routine EPI vaccinations are given at the discretion of the investigator and according to local National Plans of Immunisation schedule in each participating country. A minimum 2-week interval was to be observed between HRV vaccine and OPV doses. Of the total enrolled cohort of 60 000 subjects, 20 000 subjects were followed for efficacy and safety until one year of age while 40 000 subjects were followed for safety only until 30-90 days after the second HRV/placebo dose. A subset (N = approximately 13 000) of the 20 000 subjects are followed for efficacy and safety until 24 months of age. From the 20 000 subjects followed for efficacy and safety, a subset of 100 subjects per country (center specific, except Finland) provided two blood sample to evaluate immunogenicity.

ELIGIBILITY:
Inclusion criteria:

* Healthy infants 6-13 weeks of age at the time of the first study vaccination whose parent/guardian sign a written informed consent and whose parents/guardians can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits)

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine or placebo, or planned use during the study period
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth. (Topical steroids are allowed.)
* Child is unlikely to remain in the study area for the duration of the study
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract or other serious medical condition as determined by the investigator

Ages: 6 Weeks to 13 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63227 (Actual)
Dates: Start 2003-08-05 (Actual); Study Completion 2005-10-20 (Actual)

PRIMARY OUTCOMES:
1. Occurrence of severe RV GE caused by the wild RV strains during the period starting from 2 weeks after Dose 2 until one year of age. 2. Occurrence of definite IS cases within 31 days (Day 0 -Day 30) after each HRV vaccination dose.

SECONDARY OUTCOMES:
Severe RV GE by wild-type G1, non-G1, each non-G1, 11 score after Dose 2 and Dose 1 until 1-year old.
Severe RV GE in subset during the 2nd year and both years.
SAEs.
Definite IS until 1-year old and 2-years old.
Serum anti-RV IgA at Visits 1 and 3 (subset/country except Finland).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- GSK Investigational Site, Villanueva, Mendoza Province, Argentina
- GSK Investigational Site, Belém, Pará, Brazil
- Chile (2):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Concepción, Región Del Biobio
- GSK Investigational Site, Cali Colombia, Colombia
- GSK Investigational Site, Santo Domingo, Dominican Republic
- GSK Investigational Site, Tampere, Finland
- GSK Investigational Site, Tegucigalpa, Honduras
- Mexico (5):
  - GSK Investigational Site, Cuernavaca
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
  - GSK Investigational Site, Tlanepantla
- GSK Investigational Site, León, Nicaragua
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, Lima, Peru
- GSK Investigational Site, Valencia, Carabobo, Venezuela

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=510

REFERENCES:
- [Background] Costa Clemens SA et al. Operational organization of a large scale phase III clinical trial of rotavirus vaccine in multiple sites and countries in Latin America. Poster presented at ICP, Cancun, Mexico, 15-20 August 2004.
- [Background] De Vos B et al. Rotarix™: an effective way to prevent rotavirus diarrhoea and vomiting. Proc. 9th Congress of the Asian Pan Pacific Society of Paediatric Gastroenterology, Hepatology and Nutrition & 27th Annual Congress of the Malaysian Paediatric Association, Kuala Lumpur, 16-19 June 2005.
- [Background] Macias M et al. The rotavirus vaccine RIX4414 (Rotarix) is not associated with intussusception in one year old infants. Proc. 45th Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC), Washington DC, USA, 16-19 December 2005.
- [Background] O'Ryan et al. A novel rotavirus vaccine RIX4414 is not associated with intussusception. Proc. 44th ICAAC, Washington DC, USA, October 30-November 2, 2004.
- [Background] Ruiz-Palacios GM, Perez-Schael I, Velazquez FR, Abate H, Breuer T, Clemens SC, Cheuvart B, Espinoza F, Gillard P, Innis BL, Cervantes Y, Linhares AC, Lopez P, Macias-Parra M, Ortega-Barria E, Richardson V, Rivera-Medina DM, Rivera L, Salinas B, Pavia-Ruz N, Salmeron J, Ruttimann R, Tinoco JC, Rubio P, Nunez E, Guerrero ML, Yarzabal JP, Damaso S, Tornieporth N, Saez-Llorens X, Vergara RF, Vesikari T, Bouckenooghe A, Clemens R, De Vos B, O'Ryan M; Human Rotavirus Vaccine Study Group. Safety and efficacy of an attenuated vaccine against severe rotavirus gastroenteritis. N Engl J Med. 2006 Jan 5;354(1):11-22. doi: 10.1056/NEJMoa052434. PMID 16394298
- [Background] Vesikari et al. High efficacy of two doses of Rotarix™ (RIX4414) against rotavirus disease in Europe, Latin-America and Asia. Presented at ACPID, Cebu, Philippines, 7-10 March 2006.
- [Background] Vesikari T et al. Overcoming the safety hurdle: the rotavirus vaccine RIX4414 is not associated with intussusception. 23rd Annual Meeting of European Society for Paediatric Infectious Diseases, Valencia, Spain, 18-20 May 2005.
- [Background] Vesikari T et al. RIX4414: A new attenuated human rotavirus vaccine. 23rd Annual Meeting of European Society for Paediatric Infectious Diseases, Valencia, Spain, 18-20 May 2005.
- [Background] Buyse H, Vinals C, Karkada N, Han HH. The human rotavirus vaccine Rotarix in infants: an integrated analysis of safety and reactogenicity. Hum Vaccin Immunother. 2014;10(1):19-24. doi: 10.4161/hv.26476. Epub 2013 Oct 8. PMID 24047799
- [Background] De Vos B, Han HH, Bouckenooghe A, Debrus S, Gillard P, Ward R, Cheuvart B. Live attenuated human rotavirus vaccine, RIX4414, provides clinical protection in infants against rotavirus strains with and without shared G and P genotypes: integrated analysis of randomized controlled trials. Pediatr Infect Dis J. 2009 Apr;28(4):261-6. doi: 10.1097/INF.0b013e3181907177. PMID 19289978
- [Background] Han HH, Karkada N, Jayadeva G, Dubin G. Serologic response to porcine circovirus type 1 (PCV1) in infants vaccinated with the human rotavirus vaccine, Rotarix: A retrospective laboratory analysis. Hum Vaccin Immunother. 2017 Jan 2;13(1):237-244. doi: 10.1080/21645515.2016.1231262. PMID 27657348
- [Background] Justino MC, Araujo EC, van Doorn LJ, Oliveira CS, Gabbay YB, Mascarenhas JD, Miranda YS, Guerra Sde F, Silva VB, Linhares AC. Oral live attenuated human rotavirus vaccine (Rotarix) offers sustained high protection against severe G9P[8] rotavirus gastroenteritis during the first two years of life in Brazilian children. Mem Inst Oswaldo Cruz. 2012 Nov;107(7):846-53. doi: 10.1590/s0074-02762012000700002. PMID 23147138
- [Background] Linhares AC, Velazquez FR, Perez-Schael I, Saez-Llorens X, Abate H, Espinoza F, Lopez P, Macias-Parra M, Ortega-Barria E, Rivera-Medina DM, Rivera L, Pavia-Ruz N, Nunez E, Damaso S, Ruiz-Palacios GM, De Vos B, O'Ryan M, Gillard P, Bouckenooghe A; Human Rotavirus Vaccine Study Group. Efficacy and safety of an oral live attenuated human rotavirus vaccine against rotavirus gastroenteritis during the first 2 years of life in Latin American infants: a randomised, double-blind, placebo-controlled phase III study. Lancet. 2008 Apr 5;371(9619):1181-9. doi: 10.1016/S0140-6736(08)60524-3. PMID 18395579
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 444563/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 444563/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register